CLINICAL TRIAL: NCT00002806
Title: PHASE II STUDY OF PREIRRADIATION PCV CHEMOTHERAPY IN PATIENTS WITH SUPRATENTORIAL LOW-GRADE GLIOMAS
Brief Title: Chemotherapy Followed by Radiation Therapy in Treating Adults With Supratentorial Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-937202; CDR0000064910 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-26 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult diffuse astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma | interventions — Lomustine; Procarbazine; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- procarbazine + lomustine + vincristine + radiation (Experimental): PCV followed by external-beam cranial irradiation using at least 6 MV photons.
  Interventions: Drug: lomustine; Drug: procarbazine hydrochloride; Drug: vincristine sulfate; Radiation: low-LET photon therapy

INTERVENTIONS:
Drug: lomustine
Drug: procarbazine hydrochloride
Drug: vincristine sulfate
Radiation: low-LET photon therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining radiation therapy with chemotherapy may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of procarbazine, lomustine, and vincristine followed by radiation therapy in treating adults who have supratentorial glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Estimate the response rate of patients with newly diagnosed supratentorial low-grade glioma following neoadjuvant chemotherapy with PCV (procarbazine/lomustine/vincristine). II. Describe the toxicity of PCV. III. Determine the incidence of disease progression in these patients during PCV treatment.

OUTLINE: The following acronyms are used: CCNU Lomustine, NSC-79037 PCB Procarbazine, NSC-77213 PCV PCB/CCNU/VCR VCR Vincristine, NSC-67574 3-Drug Combination Chemotherapy Followed by Radiotherapy. PCV; followed by external-beam cranial irradiation using at least 6 MV photons.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed supratentorial * grade I/II glioma, including: Diffuse fibrillary astrocytoma No pilocytic astrocytoma No mixed tumor with ependymoma elements * Supratentorial sites include: Frontal, temporal, parietal, or occipital lobes Thalamus, basal ganglia, or midbrain Lateral or third ventricles Pons, medulla, or optic chiasm tumors allowed only if secondary to eligible tumor More than 1 separate tumor allowed Diagnosis based on surgical biopsy or subtotal resection Measurable or evaluable disease on T2-weighted MRI required

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Hematopoietic: WBC greater than 3,500/mm3 Platelet count greater than 130,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin less than 2 times upper limit of normal (ULN) AST less than 2 times ULN Alkaline phosphatase less than 2 times ULN Renal: Creatinine less than 1.5 times ULN Other: No active or uncontrolled infection No second malignancy within 3 years except: Nonmelanomatous skin cancer In situ cervical cancer No pregnant or nursing women Negative pregnancy test required within 7 days prior to entry Effective contraception required of fertile patients

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No prior chemotherapy Endocrine therapy: At least 1 week since prior steroids OR Stable steroid dose for at least 1 week prior to study Radiotherapy: No prior cranial or head and neck irradiation Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 1996-07; Primary Completion 2003-01 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Response rate | Up to 5 years

SECONDARY OUTCOMES:
Disease progression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jan C. Buckner, MD, Study Chair — Mayo Clinic
Locations (17):
- United States (17):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinical and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Background] Jenkins RB, Blair H, Ballman KV, Giannini C, Arusell RM, Law M, Flynn H, Passe S, Felten S, Brown PD, Shaw EG, Buckner JC. A t(1;19)(q10;p10) mediates the combined deletions of 1p and 19q and predicts a better prognosis of patients with oligodendroglioma. Cancer Res. 2006 Oct 15;66(20):9852-61. doi: 10.1158/0008-5472.CAN-06-1796. PMID 17047046
- [Result] Buckner JC, Gesme D Jr, O'Fallon JR, Hammack JE, Stafford S, Brown PD, Hawkins R, Scheithauer BW, Erickson BJ, Levitt R, Shaw EG, Jenkins R. Phase II trial of procarbazine, lomustine, and vincristine as initial therapy for patients with low-grade oligodendroglioma or oligoastrocytoma: efficacy and associations with chromosomal abnormalities. J Clin Oncol. 2003 Jan 15;21(2):251-5. doi: 10.1200/JCO.2003.06.023. PMID 12525516